CLINICAL TRIAL: NCT01955057
Title: Study of Psychopathological Characteristics of Patient Smoking in Thoracic Oncology
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5579
Record Dates: First submitted 2013-09-20; First posted 2013-10-07 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Smoking Cessation and Lung Cancer
MeSH Terms: conditions — Smoking Cessation; Lung Neoplasms | interventions — Thematic Apperception Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Smokers with lung cancer
  Interventions: Behavioral: Research interviews; Behavioral: Tests (Fagerström, Q-MAT, H.A.D.S, SCL 90-R); Behavioral: Projective methods (Thematic apperception Test, Rorschach); Behavioral: Carbon monoxide test

INTERVENTIONS:
Behavioral: Research interviews
Behavioral: Tests (Fagerström, Q-MAT, H.A.D.S, SCL 90-R)
Behavioral: Projective methods (Thematic apperception Test, Rorschach)
Behavioral: Carbon monoxide test

SUMMARY:
Persistent smoking after lung cancer has been the subject of medical, therapeutic and epidemiological publications for twenty years of research. Continued persistent smoking is all the more a problem for oncologists as there is evidence that smoking cessation, with lung cancer, gives therapeutic benefit. Quitting smoking can improve the response to treatments (chemotherapy, radiotherapy, surgery), quality of life and overall survival. However many patients refuse adhesion to tobacco cessation. Daily practice leads us to the hypothesis that adhesion differences aren't related to the denial of medical information, nor to resignation or to nicotine dependence. Patients who continue smoking seem to face a form of impossibility to wean. Cigarette seems to be felt as a part of their body in their narration and description of their body image.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or older
* Patient affiliated to a social security system
* Patient who has signed and dated informed consent, written before all procedures related to the study
* Patient who has received the results of the previous mandatory medical examination
* Patient who has been diagnosed with lung cancer, regardless of the histological type of the cancer
* Patient who maintains an active smoking at the time of inclusion
* Patient who has smoked at least one cigarette in the previous year of inclusion
* Patient who is being treated for lung cancer (surgery, chemotherapy, radiotherapy) and not another form of cancer
* Tobacco consumer's only by smoke inhalation
* Tobacco consumer's or tobacco associated with cannabis

Exclusion Criteria:

* Major patient under guardianship or curatorship or maintenance of justice
* Patient deprived of his liberty or in an emergency situation
* Patient with a Performance Statut(OMS) higher than 2 and/or with a psychiatric disorder like " schizophrenia and other psychotic disorders " (DSM IV)
* A palliative care patient
* Patient who began smoking during his diagnostic examination or after the diagnosis of cancer
* A pregnant or breastfeeding woman
* Patient in an exclusion period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in the pneumology ward of Strasbourg University Hospital, precisely in hospitalization units involved in cancer care (Units 1404,1403,1202,2099)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Composite indicator variable indicating the presence or absence of disturbance in one or more of the parameters evaluated: object relations, body, subject's choice. | 2 months after inclusion
  The results will be obtained:
  * From the results of each test, each has indeed a standardized rating scale
  * By analysing the content of the speech of the patient previously noted during the various interviews The investigator will classify each subject in "disturbance" or not for each of the three parameters. The presence of at least one disturbance gives the "yes" value in the indicator variable, "no" in the absence of the three disturbances.
Composite indicator variable indicating the presence or absence of disturbance in one or more of the parameters evaluated: object relations, body, subject's choice. | 4 months after inclusion
  The results will be obtained:
  * From the results of each test, each has indeed a standardized rating scale
  * By analysing the content of the speech of the patient previously noted during the various interviews The investigator will classify each subject in "disturbance" or not for each of the three parameters. The presence of at least one disturbance gives the "yes" value in the indicator variable, "no" in the absence of the three disturbances.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan GRAFFI, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Nouvel Hôpital Civil, Service de pneumologie, Unité de cancérologie thoracique, Hôpitaux Universitaires de Strasbourg, Strasbourg, France